CLINICAL TRIAL: NCT05184218
Title: A Phase 1 Study Evaluating the Safety, Tolerability, and Pharmacokinetics of Intranasal Plus Intraoral IGM-6268 in Healthy Adults and Patients With Mild to Moderate COVID-19
Brief Title: Evaluation of IGM-6268 in Healthy Adults and Patients With Mild to Moderate COVID-19
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: IGM Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: IGM-6268-002
Record Dates: First submitted 2022-01-06; First posted 2022-01-11 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2022-10

CONDITIONS: Healthy Volunteers; COVID-19
MeSH Terms: conditions — COVID-19 | interventions — IGM-6268

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to receive intranasal and intraoral administration of IGM-6268 or placebo at the assigned doses. Cohorts will be enrolled sequentially. Cohorts 1-3 and Sentinel will enroll healthy volunteers and Cohorts 4-5 and Ph1b Expansion will enroll mild-moderate COVID-19 patients.
Who Masked: Participant, Investigator
Masking Description: Double-blinded study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (7):
- Sentinel (Experimental): In the Sentinel Cohort, healthy volunteers will be randomized to receive intranasal and intraoral administration of 1 mg of IGM 6268 or placebo once per day for 5 days.
  Interventions: Drug: IGM-6268; Drug: Placebo
- Cohort 1 (Experimental): In Cohort 1, healthy volunteers will be randomized to receive intranasal and intraoral administration of 3.75 mg of IGM 6268 or placebo once per day for 5 days.
  Interventions: Drug: IGM-6268; Drug: Placebo
- Cohort 2 (Experimental): In Cohort 2, healthy volunteers will be randomized to receive intranasal and intraoral administration of 7.5 mg of IGM 6268 or placebo once per day for 5 days.
  Interventions: Drug: IGM-6268; Drug: Placebo
- Cohort 3 (Experimental): In Cohort 3, healthy volunteers will be randomized to receive intranasal and intraoral administration of 7.5 mg of IGM 6268 or placebo twice per day for 5 days.
  Interventions: Drug: IGM-6268; Drug: Placebo
- Cohort 4 (Experimental): In Cohort 4, mild-moderate Covid patients will be randomized to receive intranasal and intraoral administration of 7.5 mg of IGM 6268 or placebo once per day for 5 days.
  Interventions: Drug: IGM-6268; Drug: Placebo
- Cohort 5 (Experimental): In Cohort 5, mild-moderate Covid patients will be randomized to receive one intranasal and intraoral administration of 7.5 mg of IGM 6268 or placebo twice per day for 5 days.
  Interventions: Drug: IGM-6268; Drug: Placebo
- Ph1b Expansion (Experimental): In the Ph1b expansion cohort, mild-moderate Covid patients will be randomized to receive one intranasal and intraoral administration of 7.5 mg of IGM 6268 or placebo once or twice per day for 5 days. This cohort may be opened per Sponsor's discretion based on initial safety and activity.
  Interventions: Drug: IGM-6268; Drug: Placebo

INTERVENTIONS:
Drug: IGM-6268 — Active Comparator
Drug: Placebo — Placebo Comparator

SUMMARY:
This is a Phase 1, multi-center, randomized, double-blinded, placebo-controlled study to assess the safety, tolerability, and pharmacokinetics (PK) of IGM-6268 administered intranasally and intraorally in healthy volunteers and in outpatients with mild-moderate COVID-19. IGM-6268 or placebo will be administered by intranasal + intraoral spray using a Teleflex Mucosal Atomization Device Nasal™ Intranasal Mucosal Atomization Device once, or once or twice each day for 5 days.

DETAILED DESCRIPTION:
IGM-6268 is an engineered Immunoglobulin M (IgM) antibody that specifically targets the receptor binding domain (RBD) of the SARS-CoV-2 spike protein. This humanized pentameric IgM antibody has 10 binding sites to the spike protein and a J-chain to enable the formation of IgM pentamers.

IGM-6268 is being developed as a treatment for or prophylaxis of symptoms associated with mild to moderate COVID-19. The primary mechanism of action of IGM-6268 is to block the binding of the SARS-CoV-2 RBD on the spike protein to human angiotensin converting enzyme 2 (hACE2), the cellular receptor for SARS-CoV-2. By blocking this binding, IGM 6268 neutralizes the infectivity of the virus.

ELIGIBILITY:
Healthy Volunteers

Inclusion Criteria:

* Is male or non-pregnant female adult ≥ 18 and ≤ 55 years of age
* Has a body mass index (BMI) < 35 kg/m2.
* Is healthy as determined by medical history and physical examination
* Agrees to use contraception through 3 months after the last dose of IGM-6268

Exclusion Criteria:

* Receipt of any COVID-19 vaccine during this study and follow-up period
* Prior positive SARS-CoV2 test
* Hepatitis B virus (HBV), hepatitis C virus (HCV), or uncontrolled human immunodeficiency virus (HIV) infection
* Use of any nasally administered drug

Mild-Moderate COVID Patients

Inclusion Criteria:

* Is male or non-pregnant female adult ≥ 18 and ≤ 55 years of age
* Agrees to use contraception through 3 months after the last dose of IGM-6268
* Agrees to the collection of blood, urine, saliva, and nasopharyngeal samples, per protocol.
* Signs and symptoms of mild to moderate COVID-19 but not requiring hospitalization
* Has a laboratory-confirmed SARS-CoV-2 infection as determined by FDA-authorized antigen or NAAT diagnostic assay during the period of 72 hours prior to enrollment.

Exclusion Criteria:

* Receipt of any COVID-19 vaccine during this study and follow-up period
* Receipt of remdisivir, antiviral antibody treatment (plasma or Mabs), immosuppressive therapies, or cytokine-targeted anti-inflammatory drugs
* Concurrent use of drugs not approved for use in COVID-19 patients (e.g., ivermectin, chloroquine/hydroxychloroquine, budesonide).
* Co-morbidities including but not limited to hypertension, cardiovascular disease, diabetes (Type 1 or 2), chronic kidney disease, or asthma
* Subject is considered to be in their last few weeks of life prior to this acute illness
* Cancer within the last 5 years except stable prostate cancer and basal cell carcinoma
* Hepatitis B virus (HBV), hepatitis C virus (HCV), or uncontrolled human immunodeficiency virus (HIV) infection
* Influenza or confirmed or suspected pulmonary or systemic bacterial infection
* Receipt of any COVID-19 vaccine during this study and follow-up period
* Use of any nasally administered drug

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2022-01-20 (Actual); Primary Completion 2022-05-06 (Actual); Study Completion 2022-07-04 (Actual)

PRIMARY OUTCOMES:
Safety & tolerability of IGM-6268 by assessing the number, severity, and type of adverse events per CTCAE 5.0 | Through 60 days following receipt of final dose

SECONDARY OUTCOMES:
Concentration of IGM-6268 in serum | Predose through Day 6 (healthy volunteers) or Day 5 (mild-moderate COVID patients)
Incidence of anti-IGM-6268 antibodies in serum | Prior to dosing and at Day 28 following receipt of initial dose

CONTACTS AND LOCATIONS:
Overall Officials: Roel Funke, Study Director — IGM Biosciences, Inc.
Locations (1):
- Farmovs, Bloemfontein, Free State, South Africa